CLINICAL TRIAL: NCT06070441
Title: Adherence to Home Treatment of Patients With Neck Pain Through the Use of Information and Communication Technologies.
Brief Title: Adherence to Exercises for Neck Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, University teacher, PT, PhD, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHATBOT_NECK_PAIN
Record Dates: First submitted 2023-09-29; First posted 2023-10-06 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Treatment Adherence and Compliance
Keywords: Treatment adherence; New technologies; Back pain
MeSH Terms: conditions — Treatment Adherence and Compliance; Back Pain | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Two arms study, experimental vs control
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The interventor providing the education sessions will be blinded to group allocation The outcome assessor will be blinded to the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Home exercise assisted with a chatbot
  Interventions: Other: Education; Device: Chatbot
- Control (Active Comparator): Home exercise, usual care
  Interventions: Other: Education; Other: Home exercise, usual care

INTERVENTIONS:
Other: Education — One-week, three sessions in alternate days, outpatient supervised education on how to perform the exercises at home
Device: Chatbot — 12 week- intervention consisting of messages with an explanatory video of each exercise indicating how to do it and how many repetitions to perform
  Arms: Experimental
Other: Home exercise, usual care — 12 week- intervention. Printed sheets indicating how to exercises and how many repetitions to perform
  Arms: Control

SUMMARY:
This project continuing to study on the effectiveness of a Chatbot in promoting adherence to home physiotherapy treatment for patients, in this case, with cervical musculoskeletal injuries and pain. The use of digital technologies and media is an important option to complement in-person treatment and promote adherence to treatment at home. The research aims to verify whether the use of a Chatbot as a means of communication can produce improvements in patient adherence and clinical results.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Diagnosis of cervical pain.
* Indication of treatment through home exercises.
* With a personal smartphone
* Verbally confirms to have installed an instant messaging service or app, and accesses it at least 3 times a week

Exclusion Criteria:

* No to sign the informed consent.
* Not able to understand, read and write in the Spanish language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Adherence | 0 weeks, 12 weeks
  Record of the number of sessions performed.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | 0 weeks, 12 weeks
  Numerical scale from 0 to 10, where 0 indicates no pain and 10 is the maximum pain experienced.
Disability | 0 weeks, 12 weeks
  The Neck Disability Index (NDI) consists of ten questions in the following domains: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation. Scoring: Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability).
Satisfaction scale with the treatment received | 12 weeks
  The CRES-4 satisfaction scale consists of four items designed to evaluate whether patients are satisfied with the therapy they have received and whether it has been perceived as effective. Its global score is intended to reflect treatment effectiveness as perceived by the patient. It is a good complementary tool to judge, in particular, satisfaction with the treatment received. Consists of four questions, and score with a score ranging from 0 to 18 points. The more points, the more satisfied you are with the treatment.
Sistem usability scale | 12 weeks
  It consists of a 10 item questionnaire for measuring the usability of the experimental intervention tool with five response options for respondents, from Strongly agree to Strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, Principal Investigator — University of Valencia
Locations (1):
- David Hernández Guillén, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No